CLINICAL TRIAL: NCT01358071
Title: NGR018: Randomized Phase II Study of NGR-hTNF Plus an Anthracycline Versus an Anthracycline Alone in Platinum-resistant Ovarian Cancer
Brief Title: Phase II Study of NGR-hTNF in Combination With Doxorubicin in Platinum-resistant Ovarian Cancer
Acronym: NGR018
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGR018; 2010-023613-61 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Ovarian Cancer
Keywords: NGR-hTNF; Pegylated liposomal doxorubicin; Doxorubicin; Platinum-resistant; Progression or recurrence Ovarian Cancer; Ovarian Cancer; Advanced or metastatic
MeSH Terms: conditions — Ovarian Neoplasms; Disease Progression; Neoplasm Metastasis | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: NGR-hTNF+ anthracycline (Experimental): NGR-hTNF+Pegylated Liposomal Doxorubicin or Doxorubicin
  Interventions: Drug: NGR-hTNF; Drug: Pegylated liposomal doxorubicin; Drug: Doxorubicin
- Arm B: anthracycline (Active Comparator): Pegylated Liposomal Doxorubicin or Doxorubicin
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Doxorubicin

INTERVENTIONS:
Drug: NGR-hTNF — NGR-hTNF: 0.8 mcg/m² as 60 minutes intravenous infusion weekly or every 3 or 4 weeks until confirmed evidence of disease progression or unacceptable toxicity occurs
  Arms: Arm A: NGR-hTNF+ anthracycline
Drug: Pegylated liposomal doxorubicin — 50 mg/m² iv every 4 weeks until confirmed evidence of disease progression
Drug: Doxorubicin — 60 mg/m² iv every 3 weeks for a maximum of 8 cycles

SUMMARY:
The primary objective of this randomized phase II trial is to compare progression-free survival (PFS) in patients randomized to NGR-hTNF plus an anthracycline versus patients randomized to an anthracycline alone

DETAILED DESCRIPTION:
Considering the safety/toxicity profile of NGR-hTNF characterized by mild-to-moderate constitutional symptoms, the reversibility of these adverse events generally occurring only during the infusion time; the absence of overlapping toxicities with chemotherapeutic agents; the safety and preliminary antitumor activity observed in previous trial with doxorubicin; and the objective response rate (RR) registered in a phase II trial in previously treated ovarian cancer patients seems justified to evaluate in a randomized phase II trial the efficacy of NGR-hTNF against a doxorubicin-based option in advanced ovarian cancer patients progressing or recurrent after a standard platinum/taxane-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically-proven ovarian cancer, fallopian tube and primary peritoneal cancer in advanced or metastatic stage
* Patients previously treated with a maximum of two platinum-based regimen plus paclitaxel and with documented progressive disease on treatment (refractory patient population) or within 6 months from last chemotherapy cycle (resistant patient population)
* ECOG Performance status 0 - 2
* Life expectancy of 12 weeks or more
* Normal cardiac function
* Adequate baseline bone marrow, hepatic and renal function defined as follows:

  1. Neutrophils ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL
  2. Bilirubin ≤ 1.5 x ULN
  3. AST and/or ALT ≤ 2.5 x ULN in absence of liver metastasis or ≤ 5 x ULN in presence of liver metastasis
  4. Serum creatinine < 1.5 x ULN
* At least one (not previously irradiated) target lesion or non-measurable disease only, according to RECIST criteria
* Patients may have had prior therapy providing the following conditions are met:

  * Surgery and radiation therapy: wash-out period of 14 days
  * Systemic anti-tumor therapy: wash-out period of 21 days
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Patients must not receive any other investigational agents while on study
* More than two previous chemotherapy lines and previous treatment with anthracycline
* Patients with myocardial infarction within the last six months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Prolonged QTc interval (congenital or acquired) > 450 ms
* History or evidence upon physical examination of CNS disease unless adequately treated
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | from the date of randomization, every 6 and 8 weeks based on type of chemotherapy during treatment and every 12 weeks during the follow-up until PD or death
  Defined as the time from the date of randomization until disease progression, or death

SECONDARY OUTCOMES:
Overall survival (OS) | from the date of randomization, every 6 and 8 weeks based on type of chemotherapy during treatment and every 12 weeks during follow-up until death
  defined as the time from the date of randomization until death due to any cause.
Response Rate (RR) | from the date of randomization, every 6 and 8 weeks based on type of chemotherapy during treatment and every 12 weeks during the follow-up until PD or death
  defined as the percentage of patients who have a best-response rating of complete or partial response, according to standard RECIST criteria.
Disease Control Rate (DCR) | from the date of randomization, every 6 and 8 weeks based on type of chemotherapy during treatment and every 12 weeks during the follow-up until PD or death
  defined as the percentage of patients who have a best-response rating of complete response, partial response, or stable disease, according to standard RECIST criteria.
Duration of Disease Control | from the date of randomization, every 6 and 8 weeks based on type of chemotherapy during treatment and every 12 weeks during the follow-up until PD or death
  measured from the date of randomization until disease progression, or death due to any cause.
Safety and Toxicity according to NCI-CTCAE criteria (version 4.03) | from the start of treatment until 28 days after last treatment
  To evaluate safety and toxicity profile related to NGR-hTNF

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (8):
- Italy (6):
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione "Giovanni Pascale", Naples
  - Ospedale S. Maria della Misericordia, Perugia
  - Policlinico Universitario "Agostino Gemelli", Rome
- United Kingdom (2):
  - Beatson Oncology Centre, Gartnavel Hospital, Glasgow, Scotland
  - Clatterbridge Centre for Oncology, Bebington, Wirral